CLINICAL TRIAL: NCT04221269
Title: Post-Hospital Suicide Prevention Intervention for Patients With Schizophrenia-Spectrum Disorders
Brief Title: Suicide Prevention Intervention for Schizophrenia-Spectrum Disorders
Acronym: CLASP-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1908-001
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Suicide
Keywords: psychiatric hospitalization; suicide prevention; psychosis; psychosocial intervention
MeSH Terms: conditions — Schizophrenia; Suicide; Suicide Prevention; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment as Usual (Active Comparator): Participants assigned to Enhanced Treatment as Usual (ETAU) alone will receive unrestricted routine care in the community. Assessment feedback reports will be sent to participants' community providers at baseline, 3 months, and 6 months for care coordination.
  Interventions: Behavioral: Enhanced Treatment as Usual
- Coping Long-term with Active Suicide Program for Schizophrenia (Experimental): Coping Long-term with Active Suicide Program for Schizophrenia-Spectrum Disorders (CLASP-S) includes 3 individual sessions, 1 family meeting, and 11 phone sessions with the participant and their significant other over 6 months post-hospital discharge.
  Interventions: Behavioral: Enhanced Treatment as Usual; Behavioral: Coping Long-term with Active Suicide Program for Schizophrenia

INTERVENTIONS:
Behavioral: Enhanced Treatment as Usual — Routine community care plus assessment feedback reports to clinicians.
Behavioral: Coping Long-term with Active Suicide Program for Schizophrenia — Adjunctive psychosocial intervention for suicide prevention involving in person, family, and phone sessions.
  Arms: Coping Long-term with Active Suicide Program for Schizophrenia

SUMMARY:
The current project is a pilot randomized controlled trial to test the Coping Long-term with Active Suicide Program for schizophrenia-spectrum disorders (CLASP-S) for patients following a psychiatric hospitalization. Participants will be assigned to enhanced treatment as usual (ETAU) alone vs CLASP-S plus ETAU. Participants complete assessments at baseline during their psychiatric hospitalization and at 3 months (mid-treatment) and 6 months (post-treatment) following discharge. The primary aim is to assess the feasibility and acceptability of CLASP-S. The secondary aim is to estimate the effects of CLASP-S on reducing suicidal thoughts and behaviors relative to ETAU.

ELIGIBILITY:
Inclusion Criteria:

* suicidal thoughts or behaviors prior to hospital admission
* diagnosis of a schizophrenia-spectrum disorder
* receiving pharmacotherapy
* 18 years or older
* speaks/reads English

Exclusion Criteria:

* psychosis due to substance use or medical condition
* lack of phone access
* discharge to long-term facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 6 months
  The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score (sum of items) will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale | 6 months
  The Columbia Suicide Severity Rating Scale is an interviewer-rated measure of suicidal thoughts and behaviors. The total score (sum of items) will be used and ranges from 2 to 25 with higher scores indicating higher suicidal thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the studies published, de-identified data will be made available to other qualified researchers on request.